CLINICAL TRIAL: NCT04222868
Title: Indonesian Registry on Atrial Fibrillation
Acronym: OneAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Indonesian Heart Rhythm Society (Other)
Responsible Party: Sponsor
Other Study IDs: InaHRS-2019-001
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; registry; anticoagulant
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our rationale of creation of this registry stems from the fact that the use of VKA in patients with AF is a double-edged sword, physicians face tremendous burden in assigning patients with VKA, due to risk of Bleeding complications despite its potential benefit. We intend to seek a safe and beneficial range of INR on Indonesian patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Diagnosis of valvular or nonvalvular AF

Exclusion Criteria:

* Reversible AF
* Patients who have been enrolled as a respondent on other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study on AF registry, in which all AF patients in our hospitals that fulfilled inclusion and exclusion criteria will be input as respondents to the registry. There are two respondents for this registry, cohort, and no cohort. Noncohort registry respondents are AF patients at hospitals who fulfilled inclusion and exclusion criteria who did not consent for a 24 month follow up. Baseline characteristics of these respondents will be put to eCRF according to their hospital medical records. Patients who fulfilled inclusion and exclusion criteria who consented for a 24 month follow up were called cohort registry respondent. These respondents will be followed up at 6th, 12th and 24th month.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Adverse Cardiovascular Events | 24 months
  Major Adverse Cardiovascular Events including stroke/transient ischemic attack, thromboembolism, acute coronary syndrome
Number of Participants with Bleeding Events | 24 months
  Intracranial bleeding, gastrointestinal bleeding
Mortality Rate | 24 months
  All-cause Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sunu B Raharjo, MD, PhD, Principal Investigator — Indonesia-MoH
Locations (25):
- Indonesia (25):
  - RSUP dr. Kariadi, Semarang, Central Java
  - RSUD dr. Saiful Anwar, Malang, East Java
  - Rumah Sakit Umum Pusat Dr. M. Djamil, Padang, West Sumatra
  - RS Hasan Sadikin Bandung, Bandung
  - RS Mitra Keluarga Bekasi, Bekasi
  - RS Cirebon, Cirebon
  - RS Sanglah Denpasar, Denpasar
  - RSUPN Dr.Cipto Mangunkusumo, Jakarta
  - National Cardiovascular Center Harapan Kita, Jakarta
  - RS Bina Waluya Jakarta, Jakarta
  - RS Pasar Rebo Jakarta, Jakarta
  - RS Pusat Pertamina Jakarta, Jakarta
  - RS Siloam Kebon Jeruk Jakarta, Jakarta
  - RSPAD Gatot Subroto Jakarta, Jakarta
  - RSPAU Halim Perdanakusuma Jakarta, Jakarta
  - RSUP dr. Wahidin Sudirohusodo Makassar, Makassar
  - RSUP Prof. Dr. R. D. Kandou Manado, Manado
  - RS Adam Malik Medan, Medan
  - RS Muhammad Hoesin Palembang, Palembang
  - Eka Hospital Pekan Baru, Pekanbaru
  - RSUD Dr. Soetomo Surabaya, Surabaya
  - Eka Hospital BSD Tangerang, Tangerang
  - RS Siloam Karawaci Tangerang, Tangerang
  - RSUD Tangerang, Tangerang
  - RS Sardjito Jogjakarta, Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raharjo SB, Chandranegara AF, Hanafy DA, Yamin M, Rasyid HE, Haryadi, Rizal A, Ardhianto P, Hermanto DY, Yuniadi Y; OneAF Investigators. Indonesian registry on atrial fibrillation (OneAF). Medicine (Baltimore). 2021 May 14;100(19):e25725. doi: 10.1097/MD.0000000000025725. PMID 34106597